CLINICAL TRIAL: NCT04350047
Title: Resection of Renal Cell Carcinoma and Stage IV Inferior Vena Cava Thrombus Without Thoracotomy: A Case Series and Literature Review.
Brief Title: Renal Cell Carcinoma and Stage IV Inferior Vena Cava Thrombus: Resection Without Thoracotomy
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Parasyris, Principal Investigator, Attikon Hospital
Other Study IDs: Not appicable
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Renal Cell Carcinoma Stage III
Keywords: Renal cell carcinoma; Tumor thrombus; Inferior vena cava; level IV
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transabdominal inferior vena cava thrombectomy: Patients undergoing radical nephrectomy and inferior vena cava thrombectomy transabdominal without thoracotomy
  Interventions: Procedure: Radical nephrectomy with inferior vena cava thrombectomy without thoracotomy

INTERVENTIONS:
Procedure: Radical nephrectomy with inferior vena cava thrombectomy without thoracotomy — The abdomen was accessed through a Makuuchi incision. After mobilization of the liver and assessment of the inferior vena cava infiltration (IVC), IVC was clamped below the level of the renal veins. In order to get access to the intrapericardial IVC, an incision was made through the tendon of the diaphragm and a clamp was placed first in the hepatoduodenal ligament (Pringle maneuver) and then in the endopericardial portion of the IVC, in that order. A longitudinal 3-4 cm incision was made incorporating the junction of IVC and right renal vein. After tumor removal thrombus was removed and a fine clamp was placed at the IVC just below the hepatocaval junction and immediate release of the clamping of the hepatoduodenal ligament. Total endopericardial clamp time was 4 minutes. Patients then underwent radical nephrectomy in a standard fashion with en bloc resection of the IVC thrombus.

SUMMARY:
Assessment of short-term outcomes of radical nephrectomy combined with IVC thrombectomy with a novel technique without thoracotomy: single center case series.

DETAILED DESCRIPTION:
Assessment of the 30-day mortality and major complications as well as long-term oncological outcomes of three patients undergoing radical nephrectomy combined with inferior vena cava (IVC) thrombectomy with a novel technique without thoracotomy for renal cell carcinoma with IVC level IV thrombus. This is a retrospective case series carried out at Attikon University Hospital between January 2018 to March 2020.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Documented radiological and/or pathological diagnosis of renal cell carcinoma with level IV tumor thrombus

Exclusion Criteria:

* American Anesthesia Association (ASA) Class V and/or any contraindications to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among all patients with renal cell carcinoma operated in Attikon University Hospital, the ones with level IV tumor thrombus were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Short term mortality rate | 30 days
  Percentage of patients' postoperative deaths

SECONDARY OUTCOMES:
Short term major complications' rate | 30 days
  Incidence of Clavien/Dindo grade 3 or more postoperative complications
Recurrence rate | 27 months
  Rate of local or systemic recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Arkadopoulos, MD, PhD, Study Director — Attikon Hospital
Locations (1):
- Attikon University Hospital, Chaïdári, Greece

IPD SHARING:
Plan to Share IPD: No